CLINICAL TRIAL: NCT00553176
Title: Crohn's Therapy, Resource, Evaluation, and Assessment Tool Registry
Brief Title: The Crohn's Therapy, Resource, Evaluation, and Assessment Tool Registry
Acronym: TREAT
Status: Completed | Type: Observational
Sponsor: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR014140; WIRB® 990474 (Other: Janssen Biotech, Inc.)
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Crohn's Disease
Keywords: Infliximab; Immune disorder; Remicade; Registry; Crohn's Disease
MeSH Terms: conditions — Crohn Disease; Immune System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Crohn's disease: The Registry is an observational research program featuring clinical, economic, and humanistic measures characterizing the treatment of Crohn's disease
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — At six-month intervals (January and July), physicians will document disease characteristics, changes in Crohn's therapy, disease progression, key events, the use of ancillary services, and hospitalizations

SUMMARY:
The purpose of this study is to evaluate the long-term clinical, economic and humanistic outcomes of various treatment regimens, including infliximab, in Crohn's disease in real world medical practice.

DETAILED DESCRIPTION:
The TREAT (The Crohn's Therapy, Resource, Evaluation, and Assessment Tool) registry is a prospective, observational, multicenter, long-term registry featuring clinical, economic, and humanistic measures characterizing the treatment of Crohn's disease. The physicians will track treatments and patient outcomes over at least a 5-year period. Physicians are expected to manage patients as they would under normal practice conditions. No predefined schedule of visits or medical procedures are required. Data are collected on a semi-annual basis by physicians documenting assessment of disease severity, medication use, and adverse events. Upon enrollment, patients complete a health assessment questionnaire. As this is an observational study, no study drugs are administered. Through the course of the Registry, analyses will be performed to support submissions to health authorities, and questions of academic interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with Crohn's Disease

Exclusion Criteria:

* Patients participating in clinical trials for Crohn's disease or other conditions also were not eligible to be enrolled in the TREAT™ Registry
* Patients who are unable to participate in the program for 2 years or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with Crohn's Disease
Sampling Method: Non-Probability Sample
Enrollment: 6273 (Actual)
Dates: Start 1999-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To document the variety of treatment regimens currently employed in the management of Crohn's disease | Five years

SECONDARY OUTCOMES:
To assess clinical, economic, and humanistic outcomes of treatment | Five years
To assess the long-term impact of various Crohn's disease treatment regimens | Five years
To assess long-term outcomes specifically associated with the use of Remicade | Five years
Collection of adverse events | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Biotech, Inc. Clinical Trial, Study Director — Janssen Biotech, Inc.